CLINICAL TRIAL: NCT05733468
Title: Comparative Evaluation of Success Rate of TheraCal LC Coronal Pulpotomy and MTA Coronal Pulpotomy in Cariously Exposed Mature Permanent Molars- A Randomized Clinical Study
Brief Title: TheraCal LC Coronal Pulpotomy and MTA Coronal Pulpotomy in Mature Permanent Molars
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Dr. Vignesh R
Record Dates: First submitted 2023-02-08; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Irreversible Pulpitis; Deep Caries
Keywords: MTA; Theracal LC; Mature permanent molars; complete /coronal pulpotomy; Vital Pulp Therapy
MeSH Terms: interventions — Pemetrexed

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Theracal LC Pulpotomy (Experimental): 36 children with the cariously exposed mature permanent molar teeth indicated for pulpotomy and fulfilling the inclusion criteria will be taken for the study and coronal pulpotomy will be done till the level of root canal orifice.
  Interventions: Drug: Theracal LC
- MTA Pulpotomy (Active Comparator): 36 children with the cariously exposed mature permanent molar teeth indicated for pulpotomy and fulfilling the inclusion criteria will be taken for the study and coronal pulpotomy will be done till the level of root canal orifice.
  Interventions: Drug: MTA

INTERVENTIONS:
Drug: Theracal LC — After hemorrhage control , 1-1.5mm of TheraCal LC will be placed on the radicular pulp stumps followed by light curing, followed by the placement of IRM and composite restorative material after 2 weeks
  Other Names: Resin-modified calcium silicate
  Arms: Theracal LC Pulpotomy
Drug: MTA — After hemorrhage control , a small ball like consistency of 2-3mm of MTA will be placed on the radicular pulp stumps, followed by the placement of IRM and composite restorative material after 2 weeks
  Other Names: Bioactive calcium silicate
  Arms: MTA Pulpotomy

SUMMARY:
To evaluate and compare the clinical and radiographic success rate of TheraCal LC and MTA for coronal pulpotomy of mature permanent molar in 9-14 year children.

DETAILED DESCRIPTION:
Rationale:

Pain caused by pulpitis is one of the most common reasons for emergency dental visits. The maintenance of the vitality of the dental pulp is one of the crucial targets of modern dentistry, based on the concept of minimally invasive dentistry. Preserving the vital pulp helps in retaining proprioceptive, reparative, tooth sensitivity (innervation), vascularization, and damping functions provided by vital pulp, which help in protecting against harmful stimuli. The traditional treatment modality for permanent mature teeth with irreversible pulpitis is nonsurgical root canal treatment (NSRCT) Moreover, these treatments are lengthy and costly, and are often subject to retreatment. Many biological and clinical studies have shown that the pulp of mature teeth, which is exposed due to carious lesions, is able to be heal, and that VPT should not be limited only to young or asymptomatic teeth. Therefore, a more conservative approach of VPT has been proposed for teeth with irreversible pulpitis. A favorable outcome of this approach depends on two factors: the healing ability of the remaining vital pulp and the biocompatibility of the pulp-capping agents used. Recent studies have observed success rates ranging from 82% to 95% using modern restorative materials in mature permanent teeth, thereby suggesting that pulpotomy can be a useful alternative to RCT in adults. Hydraulic calcium silicate cements (HCSCs) are recommended as the "gold standard" material for conservative treatment of the exposed pulp. MTA is one of the most commonly used and researched material for such purposes with successful clinical outcomes. However, due to certain inherent drawbacks of MTA, such as, extended setting time and tooth discolouration there is a need for the development of newer materials to overcome the challenges associated with MTA. TheraCal LC is a material that creates a new category of resin-modified calcium silicates. It displayed significantly higher calcium-releasing ability and lower solubility than either MTA or calcium hydroxide. This high calcium release has been shown to be critical for the stimulation of apatite formation and secondary dentin bridge formation while providing a mechanical seal of the pulp. TheraCal LC doesn't discolours tooth and also have ease in handling the material with fast setting time. Hence it is been currently used in this study as pulpotomy agent to evaluate the success rate.

Aim:

To evaluate and compare the clinical and radiographic success rate of TheraCal LC and MTA for coronal pulpotomy of mature permanent molars in 9-14 year children.

Objectives :

1. To evaluate the clinical and radiographic success rate of MTA for coronal pulpotomy of mature permanent molar
2. To evaluate the clinical and radiographic success rate of TheraCal LC for coronal pulpotomy of mature permanent molar.
3. To compare the clinical and radiographic success rate of MTA and TheraCal LC for coronal pulpotomy of mature permanent molar immediate post-operative, 1 and 3 months (only clinical), 6 months and 12 months post-operative follow ups.
4. To evaluate the post-operative pain for 7 days.
5. To evaluate the correlation between the timing of hemostasis achieved and the success rate of coronal pulpotomy.

Materials and methods:

Setting: The study will be carried out in the Outpatient department of Pedodontics and Preventive Dentistry, PGIDS, Rohtak, Haryana.

Study Design: Randomized clinical study

Study Duration: This study shall be completed in a time span of 18 months.

Population: Children aged 9-14 years including both males and females diagnosed with deep carious lesion with irreversible pulpitis recruited from Outpatient department of Pedodontics and Preventive Dentistry, PGIDS, Rohtak, Haryana.

Sample size: Total number of 72 patients will be recruited in this study, with 36 patients allocated to each group

Methods: The children will be positioned supine on dental chair and examined by the dental examiners using dental chair light and mouth mirrors. Use of cotton pellets to dry the teeth and wipe away gross debris. The teeth will be anesthetized using lidocaine 2% with epinephrine 1:80000 and isolated with rubber dam. Access to the pulp chamber will be obtained after the removal of caries and exposure of the vital pulp, using a high speed bur with a water spray. Subsequently, the coronal pulp tissue will be removed down to the canal orifices. The pulp chamber will be irrigated with a light flow of water from the water syringe and excavated. A sterile cotton pellet damped in sterile saline will be placed against the pulp stumps at orifices of the root canals. The bleeding from pulp stump will be evaluated regarding the color and hemostasis achieved within 25 minutes of pressure application. After hemostasis, the test material will be placed as per the study groups.

Group 1- After hemorrhage control , 1-1.5mm of TheraCal LC will be placed on the radicular pulp stumps followed by light curing, followed by the placement of IRM cement and composite restorative material after 2 weeks following the evaluation of postoperative signs and symptoms.

Group 2- After hemorrhage control , a small ball like consistency of 2-3mm of MTA will be placed on the radicular pulp stumps, followed by the placement of IRM and composite restorative material after 2 weeks following the evaluation of postoperative signs and symptoms.

All procedures will be performed in one visit and periapical radiographs will be obtained immediately after treatment. Standardization of the X-ray will be done to have reproducibility of the X-ray during the follow-up period for evaluating the periapical changes post treatment.

Outcome measures: Clinically asymptomatic and no new periapical pathology is formed post treatment.

Statistical analysis: The data collected for each group will be entered in Microsoft excel chart to prepare a master chart. The statistical analysis for the study will be done using SPSS (Statistical Package for the Social Sciences, inc., United States). To assess the effect of independent variable on outcome variables chi square test or fischer test exact shall be utilised along with correlation and regression equation. Statistical significance will be computed and p value_< 0.05 will be considered significant.

ELIGIBILITY:
Inclusion Criteria:

1. Patient should be between 9-14 years of age
2. Intermittent or spontaneous, sharp or dull, localized, diffuse, or referred pain
3. Permanent molar tooth with deep caries and subsequent pulp bleeding evident upon excavation of caries.
4. Rapid exposure to dramatic temperature changes elicited heightened and prolonged episodes of pain even after the thermal stimulus has been removed
5. Vital bleeding pulp tissue should be present in all canals after complete pulpotomy
6. Diagnosis should be irreversible pulpitis.
7. The tooth is restorable and free from advanced periodontal disease
8. Soft tissues around the tooth are normal with no swelling or sinus tract
9. Haemostasis should be achieved after complete pulpotomy
10. The patient has non-contributory medical history

Exclusion Criteria:

1. Teeth with immature roots
2. Non-restorable
3. Pathological mobility
4. Pus discharge through an associated sinus tract
5. Swelling of associated tissues
6. Radiographic internal or external resorption or with any periapical rarefaction
7. Necrotic pulp upon exposure.
8. Bleeding beyond 25 minutes
9. Children with severe systemic illness (mental retardation/ severe psychotic disorders), prior history of allergy and any medical condition not permitting the intervention.
10. Parents and patients unwilling for participation in the study.

Ages: 9 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2024-03-01 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
Clinical success rate | Baseline to 12 months
  Clinical success criteria :
  1. No history of spontaneous pain or discomfort except for the first day after treatment
  2. No tenderness to palpation or percussion and the tooth is functional
  3. Normal mobility and probing pocket depth
  4. Soft tissues around the tooth are normal with no swelling or sinus tract
Radiographic success rate | Baseline to 12 months
  Radiographic success criteria:
  1. No pathosis evident on the radiograph such as root resorption, new furcal or periapical pathosis
  2. No canal obliteration

SECONDARY OUTCOMES:
Pain assessment | Baseline to 7 days
  To assess the intensity and incidence of pain post-operatively at every 24 hr interval for 7 days using a Visual Analog Scale (VAS) having a score from 0-10. Score 0 means no pain and score 10 means maximum pain.
Hemostasis duration | Baseline to 12 months
  To evaluate the correlation between the timing of hemostasis achieved and the success rate of coronal pulpotomy

CONTACTS AND LOCATIONS:
Overall Officials: Vignesh R, MDS, Principal Investigator — POST GRADUATE INSTITUTE OF DENTAL SCIENCES Rohtak,Haryana, India- 124001
Locations (1):
- POST GRADUATE INSTITUTE OF DENTAL SCIENCES Rohtak, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No